CLINICAL TRIAL: NCT03494998
Title: Refining and Testing the Diagnostic Accuracy of an Assessment Tool (PAT-POPS) to Predict Admission and Discharge of Children and Young People Who Attend an Emergency Department
Brief Title: Refining and Testing the Diagnostic Accuracy of PAT-POPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pennine Acute Hospitals NHS Trust (Other)
Collaborators: University Hospitals, Leicester (Other); University of Salford (Other); University of Manchester (Other)
Responsible Party: Principal Investigator, Andrew Rowland, Consultant in Paediatric Emergency Medicine, Pennine Acute Hospitals NHS Trust
Other Study IDs: 213469
Record Dates: First submitted 2018-02-26; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children and young people: Aged 0-16 years
  Interventions: Diagnostic Test: PAT-POPS

INTERVENTIONS:
Diagnostic Test: PAT-POPS — Emergency Department-specific screening tool

SUMMARY:
Increasing attendances by children (aged 0-16 years) at UK emergency departments (EDs) is putting pressure on the National Health Service (NHS). Health professionals make complex judgements on whether children attending EDs can be sent home safely or require admission. The Pennine Acute Hospitals (PAT) Paediatric Observation Priority Score (PAT-POPS) was developed as an ED-specific screening tool for this purpose. A preliminary study showed it to be a potentially effective tool for deciding admission of children from the ED. Therefore, the focus of this study is to refine the original screening tool.

ELIGIBILITY:
Inclusion Criteria:

* Children and young people aged 0-16 years of age who attend the Emergency Department

Exclusion Criteria:

* Patients who are confirmed dead on arrival at the Emergency Department
* Patients who attend the Emergency Department in cardio-respiratory arrest

Max Age: 16 Years | Sex: All
Age Groups: Child
Study Population: The study is designed in such a way that all patients, within the age range, will be enrolled into the study upon arrival at the Emergency Department. Therefore, the study population will be recruited consecutively and data collection has been planned prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Admission or discharge | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Fairfield General Hospital, Bury
  - The Royal Oldham Hospital, Oldham
  - Rochdale Infirmary, Rochdale

IPD SHARING:
Plan to Share IPD: No